CLINICAL TRIAL: NCT00490217
Title: Spontaani Bakterielli Peritoniitti: Esiintyvyys, riskitekijät ja Vaikutus Ennusteeseen
Brief Title: Spontaneous Bacterial Peritonitis: Incidence, Risk Factors and Outcome
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Other Study IDs: R065585-1
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Spontaneous Bacterial Peritonitis; Primary Peritonitis; Ascites
Keywords: Spontaneous bacterial peritonitis; incidence; Finland; etiology; liver cirrhosis
MeSH Terms: conditions — Peritonitis; Ascites; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Spontaneous bacterial peritonitis (SBP) is a severe complication of ascites in cirrhotic patients. Under clinical experience, this condition seems to be more uncommon in Finland. The aim of this study was to measure the incidence of SBP in consecutive patients with ascites requiring hospitalization in a Finnish University Hospital.

DETAILED DESCRIPTION:
Spontaneous bacterial peritonitis (SBP) is a complication of liver cirrhosis with high mortality and low survival rates. The incidence of SBP is reported to range from 11-35% in patients with ascites requiring hospitalization. Under clinical experience, the incidence of SBP in Finland seems to be lower than reported elsewhere. Alcohol is the dominant etiologic factor of liver cirrhosis in Finland (90%), which might be a factor affecting the incidence of SBP. The aim of this study is to measure the incidence of SBP in Finland. We included consecutive patients who underwent diagnostic paracentesis for ascites in Tampere University Hospital during 2/1994 - 12/1998 and 1/2005 - 3/2007. Spontaneous bacterial peritonitis was diagnosed when the ascitic fluid contained over 250 polymorphonuclear cells / mm^3 regardless of culture and with no evidence of intra-abdominal source of infection e.g. an abscess or a perforation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic paracentesis performed during the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 1993-12; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jahangir A Khan, MS, Principal Investigator — Department of Gastroenterology and Alimentary Tract Surgery, Tampere University Hospital; Pekka Collin, MD, Study Director — Department of Gastroenterology and Alimentary Tract Surgery, Tampere University Hospital; Pekka Pikkarainen, MD, Study Director — Department of Gastroenterology and Alimentary Tract Surgery, Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Pirkanmaa, Finland